CLINICAL TRIAL: NCT03597334
Title: Aerosol Therapy in Intensive Care Units: a Prospective Observation Study
Brief Title: Aerosol Therapy in Intensive Care Units
Acronym: ATICU
Status: Completed | Type: Observational
Sponsor: lvshan (Other)
Responsible Party: Sponsor-Investigator, lvshan, respiratory therapist, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PekingUPH-lvshan
Record Dates: First submitted 2018-06-19; First posted 2018-07-24 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Respiration, Artificial; Critical Care
Keywords: administration,inhalation; metered dose inhalers; nebulizers and vaporizers; bronchodilator agents; anti-bacterial agents
MeSH Terms: conditions — Respiratory Aspiration | interventions — Administration, Inhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critical ill patients: critical ill patients who admit to ICU
  Interventions: Behavioral: aerosol therapy

INTERVENTIONS:
Behavioral: aerosol therapy — Aerosol inhalation therapy refers to a local administration method in which a drug is made into aerosol particles having a very small diameter and is inhaled by a patient and the drug directly acts on the airway

SUMMARY:
Unlike in the outpatient setting, delivery of aerosols to ICU patients may be considered complex, particularly in ventilated patients. Successful delivery of aerosolized medications to ICU patients depends upon the selection of the aerosol device and its installation position, the humidification condition, and the adjustment of the ventilator mode and parameters, etc. And there is currently little guidance or information on standards of practice in aerosol therapy.

Purpose:The aim of the present work was to assess the frequency, modalities of aerosol therapy in critically ill patients either breathing spontaneously or undergoing invasive or noninvasive ventilation.

Method:This prospective cross-sectional point prevalence study will be carried out over 14 days in several intensive care units. Centers are recruited on a voluntary basis.

During the study period, characteristics of each ICU patient will be prospectively recorded each day. If patients receive inhaled medication during the study period, extensive data such as the selection of the aerosol device and its installation position will be recorded.

Data will be entered into a database and analyses will be performed using SPSS soft ware. A p value lower than 0.05 is considered signiﬁcant.

DETAILED DESCRIPTION:
Patients admitted to intensive care units (ICUs) are usually critically ill. Aerosol inhalation therapy is important for these patients. Aerosol inhalation therapy refers to a local administration method in which a drug is made into aerosol particles having a very small diameter and is inhaled by a patient and the drug directly acts on the airway. Unlike in the outpatient setting, delivery of aerosols to ICU patients may be considered complex, particularly in ventilated patients. Large particles generated by any aerosol device are trapped in the ventilator circuit and artificial airways. Moreover, the percentage of the emitted drug that is delivered past artificial airways as aerosol is lower with larger particle size. Successful delivery of aerosolized medications to ICU patients depends upon the selection of the aerosol device and its installation position, the humidification condition, and the adjustment of the ventilator mode and parameters, etc. Therefore, physicians and health-care professionals working in ICU must be adequately trained in the proper use of each aerosol device and other aerosol inhalation techniques. Otherwise, patients will receive a suboptimal dose that will not be beneficial. An international multi-center cross-sectional survey has shown that a considerable portion of aerosol inhalation therapy for patients with invasive and non-invasive ventilation need to be regulated. And there is currently little guidance or information on standards of practice in aerosol therapy. Therefore, it is necessary to carry out this study to investigate and evaluate the current clinical treatment of aerosol therapy, in order to carry out relevant education and training, and ultimately develop the standards of aerosol inhalation therapy practice in ICU.

Purpose The aim of the present work was to assess the frequency, modalities of aerosol therapy in critically ill patients either breathing spontaneously or undergoing invasive or noninvasive (NIV) ventilation.

Method This prospective cross-sectional point prevalence study will be carried out over 14 days in several intensive care units. Centers are recruited on a voluntary basis.

During the study period, characteristics of each ICU patient will be prospectively recorded each day. If patients receive inhaled medication during the study period, extensive data such as the selection of the aerosol device and its installation position will be recorded.

Data will be entered into a database and analyses will be performed using SPSS soft ware . The 95 % conﬁdence interval (CI95) of proportions are calculated for the main variables of aerosol therapy. A p value lower than 0.05 is considered signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

* patients present in intensive care unit during the study period

Exclusion Criteria:

* patients refuse to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients present in intensive care unit during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1095 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Frequency of aerosol therapy | 2 weeks
  how many aerosol therapy be administered in ICU patients

SECONDARY OUTCOMES:
drugs of aerosol therapy | 2 weeks
  the administration of atomized drugs , including type, dose, and frequency of use
Side effects of aerosol therapy | 2 weeeks
  any side effects during aerosol therapy,such as tachycardia ,hypertension,hypoxemia
selection of the aerosol device | 2 weeeks
  there are differernt types of aerosol devices which have their own characteristics.what kind of aerosol device they choose,for example pneumatic nebulizer or ultra-sonic nebulizer or vibrating mesh nebulizer or hand held devices.which is the most popullar aerosol device.
aerosol device's installation position | 2 weeeks
  For mechanical ventilated patients,position of the aerosol device in the ventilatory circuit can affect the delivery of atomized drugs.which position do practioners would choose: distal from the Y piece or inspiratory limb just before the Y piece.
humidification condition during aerosol therapy | 2 weeeks
  humidification condition can affect the delivery of atomized drugs.During aerosol therapy,how many practioner would switched off the heated humidifier

CONTACTS AND LOCATIONS:
Overall Officials: Shan Lyu, Bacelor, Principal Investigator — Peking University People's hospital ,beijing ,China
Locations (1):
- Shan Lyu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ari A. Aerosol Therapy in Pulmonary Critical Care. Respir Care. 2015 Jun;60(6):858-74; discussion 874-9. doi: 10.4187/respcare.03790. PMID 26070580
- [Background] Dhanani J, Fraser JF, Chan HK, Rello J, Cohen J, Roberts JA. Fundamentals of aerosol therapy in critical care. Crit Care. 2016 Oct 7;20(1):269. doi: 10.1186/s13054-016-1448-5. PMID 27716346
- [Background] Ari A, Harwood RJ, Sheard MM, Fink JB. Pressurized Metered-Dose Inhalers Versus Nebulizers in the Treatment of Mechanically Ventilated Subjects With Artificial Airways: An In Vitro Study. Respir Care. 2015 Nov;60(11):1570-4. doi: 10.4187/respcare.04125. Epub 2015 Jul 7. PMID 26152470
- [Background] Dugernier J, Hesse M, Vanbever R, Depoortere V, Roeseler J, Michotte JB, Laterre PF, Jamar F, Reychler G. SPECT-CT Comparison of Lung Deposition using a System combining a Vibrating-mesh Nebulizer with a Valved Holding Chamber and a Conventional Jet Nebulizer: a Randomized Cross-over Study. Pharm Res. 2017 Feb;34(2):290-300. doi: 10.1007/s11095-016-2061-7. Epub 2016 Nov 7. PMID 27822851
- [Background] Galindo-Filho VC, Ramos ME, Rattes CS, Barbosa AK, Brandao DC, Brandao SC, Fink JB, de Andrade AD. Radioaerosol Pulmonary Deposition Using Mesh and Jet Nebulizers During Noninvasive Ventilation in Healthy Subjects. Respir Care. 2015 Sep;60(9):1238-46. doi: 10.4187/respcare.03667. Epub 2015 Jun 23. PMID 26106207
- [Background] Ari A, Atalay OT, Harwood R, Sheard MM, Aljamhan EA, Fink JB. Influence of nebulizer type, position, and bias flow on aerosol drug delivery in simulated pediatric and adult lung models during mechanical ventilation. Respir Care. 2010 Jul;55(7):845-51. PMID 20587095
- [Background] Dugernier J, Wittebole X, Roeseler J, Michotte JB, Sottiaux T, Dugernier T, Laterre PF, Reychler G. Influence of inspiratory flow pattern and nebulizer position on aerosol delivery with a vibrating-mesh nebulizer during invasive mechanical ventilation: an in vitro analysis. J Aerosol Med Pulm Drug Deliv. 2015 Jun;28(3):229-36. doi: 10.1089/jamp.2014.1131. Epub 2014 Nov 13. PMID 25393556
- [Background] Lin HL, Fink JB, Zhou Y, Cheng YS. Influence of moisture accumulation in inline spacer on delivery of aerosol using metered-dose inhaler during mechanical ventilation. Respir Care. 2009 Oct;54(10):1336-41. PMID 19796413
- [Background] Ari A, Areabi H, Fink JB. Evaluation of aerosol generator devices at 3 locations in humidified and non-humidified circuits during adult mechanical ventilation. Respir Care. 2010 Jul;55(7):837-44. PMID 20587094
- [Background] Dugernier J, Reychler G, Wittebole X, Roeseler J, Depoortere V, Sottiaux T, Michotte JB, Vanbever R, Dugernier T, Goffette P, Docquier MA, Raftopoulos C, Hantson P, Jamar F, Laterre PF. Aerosol delivery with two ventilation modes during mechanical ventilation: a randomized study. Ann Intensive Care. 2016 Dec;6(1):73. doi: 10.1186/s13613-016-0169-x. Epub 2016 Jul 22. PMID 27447788
- [Background] Ehrmann S, Roche-Campo F, Bodet-Contentin L, Razazi K, Dugernier J, Trenado-Alvarez J, Donzeau A, Vermeulen F, Thevoz D, Papanikolaou M, Edelson A, Yoshido HL, Piquilloud L, Lakhal K, Lopes C, Vicent C, Desachy A, Apiou-Sbirlea G, Isabey D, Brochard L; Reva Research Network; AT@ICU Study Group. Aerosol therapy in intensive and intermediate care units: prospective observation of 2808 critically ill patients. Intensive Care Med. 2016 Feb;42(2):192-201. doi: 10.1007/s00134-015-4114-5. Epub 2015 Nov 24. PMID 26602786